CLINICAL TRIAL: NCT03601234
Title: Application of Laparoscopy Combined With Endoscopy Surgery in the Treatment of Gastric Stromal Tumors
Brief Title: Laparoscopic Endoscopic Cooperative Surgery in the Treatment of Gastric Stromal Tumors
Acronym: LECSINGST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJYFY-2017W44
Record Dates: First submitted 2018-04-25; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-04

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastric stromal tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic surgery (Experimental): This is a kind of traditional surgical method.only use laparoscopy to resect the GIST.
  Interventions: Procedure: laparoscopic surgery
- laparoscopic and endoscopic combined surgery (Experimental): LECS resects the GIST completely by laparoscopy with the help of the precise positioning and guidance of endoscopy.
  Interventions: Procedure: laparoscopic and endoscopic cooperative surgery

INTERVENTIONS:
Procedure: laparoscopic and endoscopic cooperative surgery — compare to the traditional surgery to resect the tumor,we will add the endoscopy during the operation to improve the safety and effectiveness of surgery
  Arms: laparoscopic and endoscopic combined surgery
Procedure: laparoscopic surgery — the traditional surgery
  Arms: laparoscopic surgery

SUMMARY:
Gastrointestinal stromal tumor (GIST) is a kind of mesenchymal tumor with malignant differentiation potential. It originated from mesenchymal stem cells of gastrointestinal tract.The most common is that gastric stromal tumors(GST) make up 60-70% of gastrointestinal stromal tumors.The first choice for the treatment of non-metastatic gastric stromal tumors is to ensure the integrity of the tumor and obtain the negative surgical margin.At present, the common surgical methods of resection of gastric stromal tumors include laparotomy and laparoscopy, most of them are partial gastrectomy, wedge-shaped resection, proximal subtotal gastrectomy, distal subtotal gastrectomy and total gastrectomy, etc.There was no significant difference between open surgery and laparoscopic surgery.With the rapid development of endoscopic technology in recent years, endoscopes have been continuously explored in practice.Laparoscopic endoscopic cooperative surgery(LECS) is different from the past technology. It is a new radical resection of GIST presented by Japanese scholars. LECS resects the tumor completely by laparoscopy with the help of the precise positioning and guidance of endoscopy .This method conforms to the idea of the modern minimally invasive surgery, and avoids many problems，such as incomplete resection and disorders of digestion caused by excessive tissue resection. Investigators will observe the diffenrence of LECS and traditional laparoscopic surgeries.Firstly,the investigators will collect 80 cases of GST patients, randomly assigned for the laparoscopic group, the LECS surgical treatment. Secondly, to analyzing the basic treatment and follow-up data, including the operation time, blood loss, the number of transfer laparotomy or laparoscopy, the number of cut edge positive, the distances of cut edge away from the tumor edge, the cases of anastomotic fistula bleeding, stenosis, average such confinement, the meal time, cost of treatment, tumor recurrence rate, the presence of residual stomach, upset stomach and frequency, reflux esophagitis, bile reflux gastritis and other indicators.The purpose of this subject is to observe the effectivity and safety of LECS , invent serval LECS equipment patents and provide some references for LECS applying to the minimally invasive surgery of the digestive tract tumor and multidisciplinary treatment mode.It also provides reference for gastrointestinal stromal tumors, leiomyomas, ectopic pancreas, carcinoid, early carcinomas, giant adenomas and polyps.

ELIGIBILITY:
Inclusion Criteria:

* Patients without contraindications gastroscope，surgery and anesthesia;
* Gastroscope found submucosal lesions, qualitative hard;Endoscopic ultrasonography (EUS) confirmed the lesions come from the muscularis propria;
* Tumors diameter > 2 cm;Or tumors had < 2 cm, but the position is located in the stomach wall, after nearly cardia and it is a difficult position for gastroscope ;
* Tumors diameter < 5 cm, the tumors had complete, no broken feed and bleeding;
* Not found the tumor metastasis;
* There is no history of abdominal surgery, no severe abdominal cavity adhesion
* Normal coagulation function;
* There is no history of anticoagulant drugs, or who take aspirin, salvia miltiorrhiza, etc., should stop taking drugs for more than one week;
* Patients and their families volunteered choice the surgical procedure and signed informed consent.

Exclusion Criteria:

* Patients with preoperative assessment of distant metastasis;
* Patients with preoperative radiation and chemotherapy or hormone therapy;
* Patients with acute obstruction, bleeding or perforation of the emergency surgery;
* Patients with a history of abdominal trauma or abdominal surgery;
* Patients with contraindications gastroscope，surgery and anesthesia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
operation time | 1 hours to 6 hours through the surgery completion
  record in minutes,from the beginning of anesthesia to the end

SECONDARY OUTCOMES:
blood loss | 1 hours to 6 hours through the surgery completion
  from the surgical record sheet
success rate | after the pathological report, up to 2 weeks
  to ensure the integrity of the tumor and obtain the negative surgical margin
time in bed | from two days to two weeks after surgery
  the time in bed to the postoperative patient
time to take food | from two days to two weeks after surgery
  the time to eat to the postoperative patient
postoperative complication rate | from two weeks to one year after surgery
  including anastomotic stoma fistula,anastomotic stenosis,abdominal infection,postoperative bleeding
tumor recurrence rate | from one month to two years after surgery
  periodic review the CT or MRI or endoscope
hospitalization expenses | one month
  total hospitalization expenses

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jun She, M.D; PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China